CLINICAL TRIAL: NCT04270591
Title: A Phase Ib/II, Open-Label, Multicenter Study to Evaluate the Efficacy and Safety of Glumetinib (SCC244), a Selective MET Inhibitor in Patients With Advanced Non-Small Cell Lung Cancer Harboring MET-alterations
Brief Title: Assessment of Anti-tumor and Safety in Glumetinib in Patients With c-MET-positive Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCC244-108
Record Dates: First submitted 2019-08-07; First posted 2020-02-17 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: C-Met Exon 14 Mutation
Keywords: MET; MET amplification; MET over-expression; C-Met Exon 14
MeSH Terms: interventions — glumetinib

STUDY DESIGN:
Intervention Model Description: Phase Ib：300 mg QD Glumetinib Phase II：300 mg QD Glumetinib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SCC244 300mg (Other): Phase Ib: SCC244 300mg, QD Phase II: SCC244 300mg, QD
  Interventions: Drug: Glumetinib

INTERVENTIONS:
Drug: Glumetinib — The investigational product will be orally administrated when fasting at dose level of 300mg QD
  Other Names: SCC244

SUMMARY:
Indication:Patients with Advanced c-MET-positive Non-Small Cell Lung Cancer

Phase Ib (China only):

Approximately 90 patients

Phase Ⅱ (globally):

Approximately 78 evaluable patients; addition of at least 6 patients in Safety Run-in (US only)

DETAILED DESCRIPTION:
Phase Ib study population

Approximately 90 patients with locally advanced or metastatic NSCLC (Stage IIIb, IIIc or IV) including pulmonary sarcomatoid carcinoma (PSC). All patients should carry at least one of the following MET alterations (confirmed by local or central laboratory):

* Patients with METex14 skipping mutation who had previously treated by other MET inhibitor(s)
* Patients with METex14 skipping mutation who had received 3 or more lines prior systemic therapies without MET inhibitor for the advanced NSCLC
* Patients with MET amplification (GCN ≥ 4 or MET/CEP7 ratio ≥ 2)
* Patients with MET over-expression (IHC2+) Phase II - Safety Run-in Population (US only) A minimum of 6 patients who meeting the eligibility for either Phase Ib or Phase II.

Phase II study population (globally) Approximately 78 evaluable patients with locally advanced or metastatic NSCLC (Stage IIIb, IIIc or IV, including PSC) harboring METex14 skipping mutation that have been pre-screened by local or Sponsor-designated central laboratory, who are not eligible for chemotherapy or refuse of chemotherapy after well-informed or have failed one or two prior lines of systemic therapies and have not had prior MET inhibitor for the advanced NSCLC.

ELIGIBILITY:
Inclusion criteria:

1. Provide informed consent voluntarily.
2. Male and female patients ≥ 18 years of age (or having reached the age of majority according to local laws and regulations, if the age is > 18 years).
3. Histologically or cytologically confirmed diagnosis of NSCLC including PSC.
4. Patients with stage IIIb or IIIc NSCLC who are not candidates for definitive surgical resection or concurrent chemoradiation or patients with stage IV NSCLC (AJCC version 8).
5. For Phase Ib study, patients should carry at least one of the following MET alterations (by local or Sponsor-designated central laboratory screening):

   * METex14 skipping mutation who had previously treated by other MET inhibitor(s) or
   * METex14 skipping mutation who had received 3 or more lines prior systemic therapies without MET inhibitor for the advanced NSCLC or
   * MET amplification GCN ≥ 4 or MET/CEP7 ratio ≥ 2) or
   * MET over-expression (IHC2+).
6. For Phase II study, patients with METex14 skipping mutation in tumor or ctDNA samples (local testing is acceptable for eligibility, however if the results of the central laboratory is available, the report of the central laboratory shall prevail); all patients in Phase II study will have confirmation of METex14 skipping mutation by Sponsor-designated central laboratory but this result is not necessary for eligibility.
7. Availability of tumor tissue sample (either fresh tumor biopsy or archival tumor tissue sample); for patients of phase II study (not mandatory for safety run-in), if screened and enrolled based on local test results of METex14 skipping, the tumor tissue sample must be available for central laboratory testing before C2D1; if local testing results meet the requirements, patients of phase Ib are exempt from the central laboratory confirm.
8. For Phase II study, patients are not eligible for chemotherapy or refuse chemotherapy after well-informed or have failed one or two prior lines of systemic therapies for the advanced NSCLC.

   * Treatment failure is defined as documented disease progression or intolerance to treatment.
   * Maintenance therapy given after first line chemotherapy will be considered as part of the first line if given to patients with documented response or stable disease before starting the maintenance therapy.
   * Prior neoadjuvant/adjuvant systematic therapies will count as one prior line of treatment, provided that disease recurred within 12 months of completion of neoadjuvant/adjuvant therapy.
9. For Phase II study, at least one measurable lesion as per RECIST 1.1. (A previously irradiated site lesion may only be counted as a target lesion if there is clear sign of progression since the irradiation.)
10. ECOG Performance Status (PS): 0-1.
11. Adequate bone marrow reserve, renal and liver function:

    * Absolute neutrophil count ≥ 1.5 × 109/L;
    * Hemoglobin ≥ 9 g/dL;
    * Platelet count ≥ 75 × 109/L;
    * Serum total bilirubin ≤ ULN (≤ 3 × ULN for patients with Gilbert's syndrome);
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5.0 × ULN for patients with hepatic metastasis);
    * Creatinine clearance (calculated* or measured value**) ≥ 50 mL/min

      * For calculated creatinine clearance (Ccr) value, the eligibility should be determined using the Cockcroft-Gault formula:

        * Male Ccr (mL/mim) = body weight (kg) x (140-age)/[72 x creatinine (mg/dL)]
        * Female Ccr (mL/min) = male Ccr x 0.85 ** A measured value
    * International normalized ratio (INR) < 1.3 (or < 3.0 if on anticoagulation)

Exclusion Criteria:

Patients who meet any of the following criteria shall be excluded from the study:

1. Patients with targetable activating EGFR mutation, ALK rearrangement, ROS1 rearrangement, BRAF mutation or NTRK fusion that have available standard of care therapies.
2. Patients who have symptomatic CNS metastasis which is neurologically unstable or those who have CNS disease requiring increase in the dose of steroid. (Note: Patients with controlled CNS metastasis can participate in the trial. Before entering the study, patients should have finished radiotherapy, or have received operation for CNS tumor metastasis at least two weeks before. Patients' neurological function must be in a stable state; no new neurological deficit is found during clinical examination and no new problem is found during CNS imaging examinations. If patients need to use steroids to treat CNS metastasis, the therapeutic dose of steroid should be stable for ≥ 3 months at least two weeks prior to entering the study with treatment dose no more than dexamethasone 4 mg daily or an equivalent dose of steroids.)
3. Prior exposure to MET-directed therapy (except patients harboring METex14 skipping in Phase Ib study).
4. Evidence of past or current primary malignancies other than NSCLC (except for non-melanoma skin cancer, in situ breast cancer or in situ cervical carcinoma and superficial bladder cancer, or other cancer curatively treated and with no evidence of disease for at least 5 years).
5. Subjects with clinically significant cardiovascular disease, including:

   * NYHA Class III or higher congestive heart failure;
   * History or current evidence of serious uncontrolled ventricular arrhythmias requiring drug therapy;
   * Acute myocardial infarction, severe or unstable angina pectoris, coronary artery or peripheral artery bypass graft received within 6 months prior to the first dose;
   * Left ventricular ejection fraction (LVEF) < 50%;
   * Fridericia's corrected QT interval (QTcF) > 460 ms on ECG conducted during screening;
   * Congenital long QT syndrome, or any known history of torsade de pointes (TdP), or family history of unexplained sudden death;
   * Clinically uncontrolled hypertension (after standard antihypertensive treatment, systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg);
6. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting study treatment with the exception of alopecia and grade 2 prior neuropathy.
7. Known HIV infection with a history of acquired immunodeficiency syndrome (AIDS)-defining opportunity infection within the past 12 months; active hepatitis B and hepatitis C. Patients whose test results meet one of the following will not be enrolled:

   * for patients in China and Japan, confirmed HIV antibody positive. For patients in the US, patients with a history of HIV but no history of AIDS or an AIDS-defining opportunistic infection are allowed to be enrolled;
   * serum HBsAg positive and HBV DNA>200 IU/ml or 1000 copies/mL;

     - For patients in Japan, whose results are HBsAg antigen negative; however, when HBsAb or HBcAb positive, the patients whose HBV DNA < 200 IU/ml or 1000 copies/mL could be enrolled.
   * serum HCV antibody and HCV RNA positive.
8. Anticancer therapy (including chemotherapy, targeted therapy, biotherapy, hormone therapy or other investigational agents) within 4 weeks or 5 times of half-lives (whichever is shorter) prior to the first dose of the study drug or who have not recovered from the side effect of such therapy.
9. Radical radiation therapy (including radiation therapy for over 25% bone marrow) within 4 weeks prior to the first dose of the investigational product or received local palliative radiation therapy for bone metastases within 2 weeks.
10. Major surgery or had significant traumatic injury within 28 days prior to the first dose of the investigational product.
11. Patients who have to receive treatment (definite strong CYP3A4 inhibitor or inducer [appendix 6]; in addition, herbals/supplements containing St. John's wart [Hypericum perforatum L.] and Sevillia orange etc. should also be avoided.) that is prohibited during the study and those who cannot discontinue drugs (e.g. antiarrhythmic agent) that may lead to QTc interval prolongation or torsade de pointes. Additionally, patients who have to receive treatment of strong inhibitor for CYP2C8 and/or CYP2C9 [appendix 6] and substrates or inhibitor for transporter [appendix 7] will be excluded in safety run-in part of the study.
12. Any diseases or medical conditions, at the investigator's discretion, that may be unstable or influence their safety or study compliance, including organ transplantation, abuse of psychotropic medication, alcohol abuse or history of drug abuse.
13. Other serious illness or medical conditions at the investigator's discretion, that may influence study results, including but not limited to serious infection, diabetes, cardiovascular and cerebrovascular diseases or lung disease.
14. Patients with a history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment or any evidence of clinically active ILD.
15. Pregnant or breast-feeding patients. Pregnancy refers to the state of a woman between fertilization and the end of pregnancy confirmed by positive laboratory hCG test (> 5 mIU/mL). Breast-feeding woman can become eligible for this study if she stops breast-feeding, however, cannot restart the breast-feeding on/after the completion of the study treatment.
16. Man and woman with childbearing potential (WOCBP refer to appendix 3) not using effective contraception (refer to appendix 3) during the trial and within 6 months after the end of treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2023-10-25 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | through study completion, an average of 1 year
  ORR as determined by an Independent Radiology Review Committee (IRRC) according to RECIST Version 1.1.

SECONDARY OUTCOMES:
ORR(assessed as per investigators) | through study completion, an average of 1 year
  ORR (assessed as per investigators)
DOR | The time from the date of first documented partial response or complete response to progressive disease or death, an average of 6 months
  DOR
Efficacy of glumetinib | Through study completion, an average of 1 year.
  OS

CONTACTS AND LOCATIONS:
Overall Officials: James Zhou, MD, Study Director — Haihe Biopharma
Locations (44):
- United States (2):
  - Norton Cancer Institute, Louisville, Kentucky
  - The Oncology Institute of Hope & Innovation, Louisville, Kentucky
- China (31):
  - Anhui Province Hospital, Hefei, Anhui
  - The Chest Hospital of Anhui Province, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospita, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Union Medical College Hospital Affiliated to Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Cancer Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Hainan Cancer Hospital, Haikou, Hainan
  - Cancer Hospital Affiliated to Harbin Medical University, Harbin, Heilongjiang
  - Henan Province Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Wuhan Union Hospital, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province People's Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Affiliated Hospital of Hebei University, Baoding, Shandong
  - Shandong University Qilu Hospital, Jinan, Shandong
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Fudan university Shanghai cancer center, Shanghai, Shanghai Municipality
  - The Chest Hospital of Shanghai, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital，College of of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Province Cancer Hospital, Hangzhou, Zhejiang
  - Hunan Province Cancer Hospital, Changsha
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Japan (11):
  - Ehime University Hospital, Ehime
  - Kyushu University Hospital, Fukuoka
  - Kanagawa Cancer Center, Kanagawa
  - Niigata Cancer Center Hospital, Niigata
  - Kindai University Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Hokkaido University Hospital, Sapporo
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital East, Tokyo
  - National Cancer center, Tokyo
  - Tottori University Hospital, Tottori

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Background] Drilon AE CD, Ou S-H. Efficacy and safety of crizotinib in patients (pts) with dvanced MET exon 14-altered non-small cell lung cancer (NSCLC). J Clin Oncol. 2016; 34:suppl; abstr 108.
- [Background] 6. Felip E HL, Patel JD. Tepotinib in patients with advanced non-small cell lung cancer harboring MET exon 14-skipping mutations: Phase II trial. . J Clin Oncol. 2018; 36:suppl; abstr 9016.
- [Background] Yin L, Lu Y. [MET Exon 14 Skipping Mutations in Non-small Cell Lung Cancer]. Zhongguo Fei Ai Za Zhi. 2018 Jul 20;21(7):553-559. doi: 10.3779/j.issn.1009-3419.2018.07.09. Chinese. PMID 30037377
- [Background] Vuong HG, Ho ATN, Altibi AMA, Nakazawa T, Katoh R, Kondo T. Clinicopathological implications of MET exon 14 mutations in non-small cell lung cancer - A systematic review and meta-analysis. Lung Cancer. 2018 Sep;123:76-82. doi: 10.1016/j.lungcan.2018.07.006. Epub 2018 Jul 6. PMID 30089599
- [Background] Liu SY, Gou LY, Li AN, Lou NN, Gao HF, Su J, Yang JJ, Zhang XC, Shao Y, Dong ZY, Zhou Q, Zhong WZ, Wu YL. The Unique Characteristics of MET Exon 14 Mutation in Chinese Patients with NSCLC. J Thorac Oncol. 2016 Sep;11(9):1503-10. doi: 10.1016/j.jtho.2016.05.016. Epub 2016 May 30. PMID 27257131
- [Background] Frampton GM, Ali SM, Rosenzweig M, Chmielecki J, Lu X, Bauer TM, Akimov M, Bufill JA, Lee C, Jentz D, Hoover R, Ou SH, Salgia R, Brennan T, Chalmers ZR, Jaeger S, Huang A, Elvin JA, Erlich R, Fichtenholtz A, Gowen KA, Greenbowe J, Johnson A, Khaira D, McMahon C, Sanford EM, Roels S, White J, Greshock J, Schlegel R, Lipson D, Yelensky R, Morosini D, Ross JS, Collisson E, Peters M, Stephens PJ, Miller VA. Activation of MET via diverse exon 14 splicing alterations occurs in multiple tumor types and confers clinical sensitivity to MET inhibitors. Cancer Discov. 2015 Aug;5(8):850-9. doi: 10.1158/2159-8290.CD-15-0285. Epub 2015 May 13. PMID 25971938
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Result] Jemal A, Siegel R, Xu J, Ward E. Cancer statistics, 2010. CA Cancer J Clin. 2010 Sep-Oct;60(5):277-300. doi: 10.3322/caac.20073. Epub 2010 Jul 7. PMID 20610543
- [Derived] Lu S, Yu Y, Zhou J, Li X, Goto K, Min X, Nishino K, Cui J, Wu L, Sakakibara J, Shu Y, Dong X, Li L, Yoneshima Y, Zhou C, Li X, Zhang Y, Huang D, Zang A, Zhang W, Wang X, Zhang L, Bai C, Fang J, Cao L, Zhao Y, Yu Y, Shi M, Zhong D, Li F, Duanmu W, Wang Y. Long-term follow-up results from the GLORY study: phase II study of gumarontinib in East Asian patients with MET exon 14 skipping mutated non-small cell lung cancer. Transl Lung Cancer Res. 2025 Sep 30;14(9):3924-3938. doi: 10.21037/tlcr-2025-638. Epub 2025 Sep 28. PMID 41132955
- [Derived] Yu Y, Dong W, Shi Y, Wu R, Yu Q, Ye F, Zhou C, Dong X, Li X, Li Y, Li Z, Wu L, Pan Y, Shen H, Wu D, Xu Z, Wu J, Xu N, Qin Y, Zang A, Zhang J, Zhou J, Zhang X, Zhao Y, Li F, Wang H, Liu Q, Han Z, Li J, Lu S. A pooled analysis of clinical outcome in driver-gene negative non-small cell lung cancer patients with MET overexpression treated with gumarontinib. Ther Adv Med Oncol. 2024 Jul 31;16:17588359241264730. doi: 10.1177/17588359241264730. eCollection 2024. PMID 39091606
- [Derived] Yu Y, Zhou J, Li X, Goto K, Min X, Nishino K, Cui J, Wu L, Sakakibara J, Shu Y, Dong X, Li L, Yoneshima Y, Zhou C, Li X, Zhang Y, Huang D, Zang A, Zhang W, Wang X, Zhang L, Bai C, Fang J, Cao L, Zhao Y, Yu Y, Shi M, Zhong D, Li F, Li M, Wu Q, Zhou J, Sun M, Lu S. Gumarontinib in patients with non-small-cell lung cancer harbouring MET exon 14 skipping mutations: a multicentre, single-arm, open-label, phase 1b/2 trial. EClinicalMedicine. 2023 Apr 6;59:101952. doi: 10.1016/j.eclinm.2023.101952. eCollection 2023 May. PMID 37096188